CLINICAL TRIAL: NCT00211055
Title: A Multicenter, Epidemiological, Observational Study of the Management of Anemia in Critically Ill Pediatric Patients
Brief Title: A Study to Observe the Causes and Treatment of Anemia in Critically Ill Children
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Other Study IDs: CR004396
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Anemia
Keywords: Critically Ill; Intensive Care Unit; Blood transfusion; Blood loss; Pediatric; Children; Anemia, Pediatric Intensive Care Unit; Hemoglobin; Transfusion
MeSH Terms: conditions — Anemia; Critical Illness; Hemorrhage

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine the incidence of anemia and blood transfusions and management of these in critically ill children

DETAILED DESCRIPTION:
Critically ill patients admitted to the intensive care unit often have anemia from one or more of a number of possible causes including blood loss due to surgery or injury, frequent blood sampling, chronic diseases such as kidney failure or cancer or treatments being received, such as chemotherapy. Although the common treatment for anemia is red blood cell transfusion, the current guidelines for blood transfusions for children are based on available information regarding transfusions in adults. Since many characteristics specific to critically ill children may affect the way in which they respond to anemia and transfusion, additional information is needed to better define guidelines for the prevention and treatment of anemia in critically ill children. This is a multi-center study to collect information regarding the management of anemia in critically ill children. Information needed to evaluate anemia, blood loss and transfusions will be collected from the patients' hospital records. No blood draws or procedures will be required by this survey and no medication will be supplied by the study Sponsor. Each patient's treating physician will be responsible for all decisions regarding his/her clinical care and treatment during the study. Approximately 1200 patients will be enrolled into this study, which is divided into 2 parts. During part 1, at least 400 patients who are newly admitted to the Pediatric Intensive Care Unit (PICU) will be enrolled, regardless of their length of stay in the PICU. During part 2, up to an additional 800 patients who are newly admitted into the PICU and have remained there for > = 48 hours at the time of entry into the study will be enrolled. Information for each patient will be collected for up to 28 days or until time of discharge from the hospital or death of the patient, whichever occurs first. Blood loss will be reported for each day the patient remains in the PICU; information regarding the treatment of anemia, including number and reasons for transfusions will be collected for a maximum of 28 days, regardless of the length of stay in the PICU. Information collected at the time of discharge from the hospital will include date of discharge and whether or not the patient is receiving mechanical assistance to breathe. Several possible hypotheses are being generated in this study: 1) Blood loss due to procedures and routine laboratory tests may be a major cause of anemia and transfusions in critically ill children; 2) Determining significant causes of anemia and blood transfusions in children will allow for better future treatment of anemia; and 3) Pediatric patients who receive blood transfusions have more days on a ventilator (a machine that helps patients who cannot breathe on their own), longer stays in the PICU and decreased organ function. Since the study involves only collection of information, no treatment will be required by the Sponsor and no medication will be supplied by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 0 to 17 years
* During part 1 of this study, patients must be newly admitted to the Pediatric Intensive Care Unit (PICU) (regardless of stay)
* During part 2 of the study, patients must be newly admitted to the PICU and have stayed there for > = 48 hours
* Patients' legally acceptable representatives must have signed an informed consent
* Patients aged 7 years and above must give assent if or when they are physically capable

Exclusion Criteria:

* Premature infants (patients who were born at < = 37 weeks who are < 28 days old)
* Patients who have previously participated in this study
* Patients from a family unwilling to receive blood transfusions (for example for religious reasons)
* Patients who are participating in any other transfusion or blood-related research at the time of entry into the study or any time during the study
* Patients who are known to be pregnant (no pregnancy test will be performed in this study)
* Patients with known or suspected brain death
* Patients who have had a Pediatric Intensive Care Unit (PICU) stay of longer than 72 hours within the 7 days prior to entering the study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1201 (Actual)
Dates: Start 2004-09; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.